CLINICAL TRIAL: NCT05605769
Title: Evaluation of the Performance of Rapid Diagnostics for SARS-CoV-2 Self-testing in the Hands of Untrained Users
Brief Title: Evaluation of the Performance of Rapid Diagnostics for SARS-CoV-2 Self-testing in the Hands of Untrained
Acronym: CV009
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: CV009
Record Dates: First submitted 2022-10-31; First posted 2022-11-04 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: COVID-19
Keywords: Covid 19 self- testing, lay users
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to independently evaluate the usability and performance of rapid assays detecting SARS-CoV-2 antigen(s) and intended for self-testing. For this, the results of the test performed and interpreted by an untrained lay user will be compared to the results obtained by a trained healthcare professional using the same test kit, and, separately, to the current gold standard for testing, RT-PCR detecting SARS-CoV-2 RNA

DETAILED DESCRIPTION:
The COVID-19 pandemic has rapidly spread across the globe. As 03 March 2022, there are approximately 438 517 285 confirmed cases worldwide. Recent surge of new infections globally due to omicron variant led to significant increase of testing demand. Although rapid diagnostic tests (RDT) detecting SARS-CoV-2 antigens are now authorized in most countries and contribute substantially to expanding of testing capacity, shortage of healthcare resources is an important barrier to further scale up. Self-testing has been widely used in many high-income countries as an additional tool to provide convenient and timely access to testing. A number of self-tests detecting SARS-CoV-2 have been authorized by stringent regulatory authorities (SRA) such as US Food and Drug Administration (FDA), CE-IVD, Health Canada, Therapeutics Goods Administration (TGA) under an Emergency Use Authorization (EUA). In low- and middle-income countries (LMIC) self-testing for SARS-CoV-2 has not yet been widely adopted. Data on self-test use in LMIC are still very limited and the performance of SARS-CoV-2 self-test assays was not evaluated in LMIC settings. Additionally, the price for self-test kits is often prohibitive to its wide use in low resource settings. In 2021, FIND, the Diagnostic Alliance, through an open request for proposal (RFP) has identified several manufacturers of affordable and easy-to-use self-testing assays for SARS-CoV-2 antigen detection in nasal swabs and saliva specimens. FIND and [NAME OF THE PARTNER] aim to evaluate these novel affordable self-testing solutions in LMIC settings in a 2-phase study

ELIGIBILITY:
Phase 1 Inclusion Criteria:

* 18 years of age
* Able to speak and read local language depending on site of recruitment
* Provided voluntary written consent to participate in this stud

Phase 11 inclusion Criteria:

* 18 years of age
* Able to speak and read local language depending on site of recruitment
* Suspected to have COVID-19 (as per WHO or national guidelines).
* SYMPTOMATIC group)
* Contacts of confirmed cases of COVID-19
* Individuals residing or working in an area with high risk of transmission of virus
* Individuals residing or travelling to an area with community transmission
* Individuals working in any health care setting, including within health facilities or within the community
* Written consent
* Provided the required number of specimens suitable for testing. Exclusion criteria
* Participated in Phase I or Phase II of the study
* Prior medical or clinical laboratory training
* Prior experience with self-testing for SARS-CoV-2
* Hemodynamic instability as determined by the treating physician
* unable to cooperate with respiratory sample collection or on oxygen therapy
* Recent history of excessive nose bleeds
* Any condition which, in the opinion of the investigator feels unable to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants from general population who are able to read the local language and have no prior experience with covid self-specimen collection and testing. For Phase II, (less than 18 years) old suspected to be infected with SARS-CoV-2 (as per national or WHO guidelines) presenting at the testing site(s) will be invited to participate.
  Participants will come from the following countries: Georgia, South Africa, Uganda and Peru
Sampling Method: Non-Probability Sample
Enrollment: 3266 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
To determine the SARS-CoV-2 self-tests label comprehension by the intended users by assessing the extent to which the users understand the information in the self-test labelling | 4 weeks
  Proportion of study participants that correctly comprehend key messages from packaging and labelling measured by the proportion of participants providing correct responses to a self-administered semi-structured question
To determine the ability of the intended users to correctly interpret testing results by evaluating the correctness of user's interpretation of contrived results | 4 weeks
  Percentage of the agreement between the pre-defined results of contrived self-testing devices and their interpretation by study participants
Phase 11 Outcomes | 6weeks
  a. Proportion of participants that performed the self-testing procedure correctly and usability index of each testing step (Proportion of participants that performed each step correctly); documented errors and difficulties faced at each self-testing step

SECONDARY OUTCOMES:
To evaluate the usability in specific subgroups defined based on demographic characteristics such as age and education level | 6 weeks
  Proportion of participants that correctly comprehend key messages from packaging and labelling, performed the self-testing procedure and interpreted the results correctly in specific subgroups defined based on age and educational level. Documented errors and difficulties at each self-testing step in these subgroups
To evaluate diagnostic accuracy of SARS-CoV-2 self-tests in specific subgroups defined based on the presence of symptoms, RT-PCR Ct values, vaccination status | 6 weeks
  Point estimates of sensitivity and specificity of index test with 95% confidence intervals in specific subgroups defined based on presence of symptoms, RT-PCR Ct values, vaccination status

CONTACTS AND LOCATIONS:
Overall Officials: Maia Alkhazashvili, MD, Principal Investigator — Lugar Centre; Isaac Ssewanyana, Phd, Principal Investigator — Uganda National Laboratory Services; Mohhamed Majam, Msc, Principal Investigator — Ezintsha Research Centre; Cesar Ugarte, Phd, Principal Investigator — UPCH
Locations (2):
- Ezintsha Research Centre, Johannesburg, Guateng, South Africa
- Uganda National Health Laboratories Services, Kampala, Uganda